CLINICAL TRIAL: NCT01894646
Title: PET Imaging of Extrathalamic α4β2-nicotinic Acetylcholine Receptors in Health and Disease With [18F]XTRA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We terminated the study due to lack of funding
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00076249; 1R21AG037298-01A1 (NIH)
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Measure of Uptake of XTRA in the Brain
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Young healthy individuals (ages 18-50) (Experimental): Positron Emission Tomography (PET) Imaging
  Interventions: Radiation: Positron Emission Tomography (PET) Imaging
- Elderly healthy individuals (ages 60-85) (Experimental): Positron Emission Tomography (PET) Imaging
  Interventions: Radiation: Positron Emission Tomography (PET) Imaging
- Patients with Alzheimer's disease or mild cognitive impairment (Other): Positron Emission Tomography (PET) Imaging
  Interventions: Radiation: Positron Emission Tomography (PET) Imaging

INTERVENTIONS:
Radiation: Positron Emission Tomography (PET) Imaging

SUMMARY:
Currently, only three radiotracers, (2-[18F]FA, 6-[18F]FA and [18F]AZAN), are available for studying α4β2-nicotinic acetylcholine receptors (α4β2-nAChR) in human brain using PET imaging. A crucial problem for 2-[18F] FA, 6-[18F] FA and ([18F] AZAN is low binding potential (BP) in extrathalamic (ET) regions, including hippocampus, cortex and caudate which have lower receptor densities than the thalamus. The importance of imaging ET-α4β2-nAChRs (ET-nAChR) has emerged from the post-mortem demonstration of altered densities of ET-nAChRs (but not thalamic nAChR) in neurodegenerative diseases and schizophrenia. PET imaging of ET-nAChR may prove to be useful in both detecting early changes and following functional deterioration in neurodegenerative diseases such as Alzheimers disease. Furthermore, PET imaging of ET-nAChR may allow investigation and development of new therapies acting on the acetylcholine system.

The imaging drawbacks of the presently available nAChR radioligands have initiated the development of radioligands with greater binding potential by several research groups. The available pre-clinical data on the investigators' new radioligand [18F](-)-JHU86428 ([18F]XTRA) suggest that this radioligand is superior to 2-[18F]FA for quantitative PET imaging of α4β2-nAChR (Gao, J. Med. Chem, 2008). In baboon PET studies [18F]XTRA exhibits 200% greater brain uptake, 300% higher BPs and reaches steady-state in approximately 1.5 h in cortical regions post-bolus administration versus 6-8 h for 2-[18F]FA. In vitro binding assays shows greater binding affinity of XTRA and similar nAChR-subtype selectivity in comparison with 2-FA. Both ligands bind selectively with the β2-subtypes that are predominant nAChR subtypes in the mammal brain and display little binding affinity at ganglionic α3β4-nAChR.

The current planned human protocol will be conducted to (1) determine brain distribution (brain uptake) and test the reproducibility (in test-retest design) of [18F]XTRA brain PET scans for validation of the radioligand; (2) generate estimates of the whole body and internal organ radiation absorbed doses from exposure to single iv administrations of [18F]XTRA in healthy human subjects; and (3) determine brain distribution of [18F]XTRA in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

The population consists of healthy adults 18-85 years of age. There is no race or sex bias in our recruitment.

a. Inclusion criteria.

1. healthy volunteer, 18-80 years of age, and in portion 2, patient with Alzheimer's disease or patient with mild cognitive impairment (age 60-80 years)
2. screening laboratory tests will be obtained for subjects within a 10-day period prior to the PET study and the results must be within normal limits for gender and age. These tests will be repeated with a 10-day window following the PET study.
3. ECG conducted within a 10-day period prior to the PET study. The ECG will be repeated within 10 days following the study.
4. No contraindications to MRI scanning if MRI is to be obtained in the section for which the subject participates. These contraindications include pacemakers, metallic implants/prosthesis or prohibitive claustrophobia, etc.
5. No contraindications to PET scanning to include pregnancy, etc. For females of childbearing potential, negative serum pregnancy test obtained within a 10-day period prior to PET study
6. Subject agrees to return to the Hospital for f/u ECG and laboratory testing of blood and urine

Exclusion Criteria:

1. Participants with history of epilepsy, focal structural CNS abnormality such as stroke, or arteriovenous malformation
2. History of head injury with loss of consciousness > 1 hour,
3. Active substance abuse (drugs or alcohol) or active nicotine use
4. ECG demonstrating the participant is not in a sinus rhythm or is having acute ischemia
5. Any medical condition that in the opinion of the study investigators would constitute a safety risk to the subject.
6. Any radiation exposure in the past calendar year that in combination with the radiation exposure from this study would exceed 5 rem

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
PET Imaging of extrathalamic α4β2-nicotinic acetylcholine receptors in health and disease with [18F]XTRA | 1 year
  Measures brain uptake of F18 XTRA

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States